CLINICAL TRIAL: NCT02048787
Title: An Open-label, Single Dose, Multicenter Study to Evaluate the Pharmacokinetics and Safety of 50 mg Oral Buparlisib in Subjects With Moderate and Severe Renal Impairment Compared to Matched Control Healthy Volunteers.
Brief Title: Pharmacokinetic Study of Buparlisib in Subjects With Renal Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CBKM120C2113; 2013-003384-64 (EudraCT Number)
Record Dates: First submitted 2014-01-20; First posted 2014-01-29 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2015-12

CONDITIONS: Renal Impairment
Keywords: Renal impairment; Healthy volunteers; Clinical pharmacology study
MeSH Terms: conditions — Renal Insufficiency | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate renal impairment group (Experimental): Subjects with moderate renal impairment defined as eGFR of 30-59 mL/min/1.73m2 at screening can be enrolled in this group
  Interventions: Drug: Buparlisib
- Severe renal impairment group (Experimental): Subjects with severe renal impairment defined as eGFR of 15-29 mL/min/1.73m2 at screening can be enrolled in this group
  Interventions: Drug: Buparlisib
- Matching healthy control group (Experimental): Subjects with normal renal function defined as eGFR ≥ 90 mL/min/1.73m2 at screening and matching to the renal impaired subject based on gender, race, age, and weight can be enrolled in this group.
  Interventions: Drug: Buparlisib

INTERVENTIONS:
Drug: Buparlisib — Subjects will receive a single dose of 50 mg buparlisib.
  Other Names: BKM120

SUMMARY:
To characterize the pharmacokinetics and safety of buparlisib following a single 50 mg oral dose in subjects with moderate and severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Other than renal impairment, subjects should be in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, (except for additional inclusion criteria for renal impaired patients).
* Subjects must have a BMI between 18 kg/m2 and 34 kg/m2 and weight at least 50 kg and no more than 120 kg.

  * Additional criteria for renal impaired subjects: - Subjects must have stable renal disease without evidence of renal progressive disease defined as moderate renal impairment (eGFR 30-59 mL/min/1.73m2) or severe renal impairment (eGFR 15-29 mL/min/1.73m2).
  * Additional criteria for matched healthy control subjects: - Matched to at least one renal impaired subject by gender, race, age (± 10 years), and weight (± 20%).
* An estimated GFR as determined by MDRD equation within normal range as determined by eGFR ≥ 90 mL/min/1.73m2

Exclusion Criteria:

* Significant illness, including infections, or hospitalization within the 2 weeks prior to dosing, except for the renal impaired subjects who due to their renal disease may be affected by significant medical problems which require frequent hospitalizations.
* Any surgical or medical condition that may significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study
* Subject has a medical history of cardiac disease and/or clinically significant ECG abnormalities within 6 months prior to screening.
* Subject has an active or a history within 6 months prior to screening of clinically significant hematologic, endocrinologic, pulmonary, cardiovascular, hepatic, or allergic disease, medically documented (other than clinical conditions associated with renal impairment for the renal impaired subjects only).
* - Additional exclusion criteria for renal impaired subjects: - Severe albuminuria > 300 mg/day.
* Subjects undergoing any method of dialysis.
* Subjects with renal impairment due to hepatic disease (hepatorenal syndrome).
* Subjects with clinically significant abnormal findings, not consistent with clinical disease, upon physical examination, ECG or laboratory evaluation.
* Use of any prescription or non-prescription medication that has the potential to interact with buparlisib within two weeks prior to dosing or during the study.
* - Additional criteria for matched healthy control subjects: - Use of any prescription or non-prescription medication or vitamins during 14 days prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter Cmax | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the maximum plasma concentration (PK parameter Cmax). Cmax directly determined from the plasma concentration-time profiles.
Plasma PK parameter AUCinf | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter AUCinf (area under the plasma concentration-time curve from time 0 to infinity). AUC determined from the plasma concentration-time profile using non-compartmental analysis.
Plasma PK parameter AUC0-t | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter AU0-t (area under the plasma-concentration time curve from timepoint 0 to time t). AUC determined from the plasma concentration-time profile using non-compartmental analysis.
Plasma PK parameter CL/F | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter CL/F (clearance).
Urine PK parameter CLR | predose, 0-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, 120-144 h
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the urine clearance CLR.

SECONDARY OUTCOMES:
Plasma PK parameter Tmax | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter Tmax (time to reach maximum plasma concentration), directly determined from the plasma concentration-time profile.
Plasma PK parameter T1/2 | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter T1/2 (terminal half-life).
Plasma PK parameter Vz/F | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter Vz/F (the apparent volume of distribution following extravascular administration).
Plasma Protein Binding | predose, 1 hour post-dose
  Measurement of effect of renal impairment on plasma protein binding. Fraction of buparlisib unbound will be determined (Fu).
Unbound plasma PK parameter Cmax,u | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter Cmax,u (Cmax,u is the observed maximum unbound plasma concentration following administration).
Unbound plasma PK parameter AUCinf,u | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameters AUCinf,u (AUCinf,u is the area under the unbound plasma concentration-time curve extrapolated to infinity).
Unbound plasma PK parameter Vu/F | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter Vu/F (the apparent unbound drug volume of distribution following extravascular administration).
Unbound plasma PK parameter CLu/F | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameter CLu/F (the unbound systemic clearance from plasma).
Urine PK parameter Ae0-t | predose, 0-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h, 48-72 h, 72-96 h, 96-120 h, 120-144 h
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the urine PK parameter Ae0-t (the amount of unchanged buparlisib excreted into the urine from time 0 to a defined point in time).
Relationship between PK parameters Cmax, AUCinf, AUC0-t, CL/F, urine CLR and renal function. | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Determination of the relationship between the primary PK parameters (Cmax, AUCinf, AUC0-t, CL/F and urine PK parameter CLR) and renal function parameters eGFR (estimated glomerular filtration rate using the equation from the Modification of Diet in Renal Disease (MDRD) study).
Adverse Events severity and frequency | Baseline Day 1 to 30 days post-dose
  Assessment of safety and tolerability of a single dose buparlisib in renal impaired subjects compared with healthy control subjects by assessing the frequency and severity of Adverse Events based on the CTCAE criteria.
Change from baseline in laboratory parameters | From baseline Day 1 to 30 days post-dose
  Assessment of safety and tolerability of a single dose buparlisib in renal impaired subjects compared with healthy control subjects by assessing the change from baseline in hematological and biochemical laboratory parameters.
Change from baseline in ECG parameters | From baseline Day 1 to 30 days post-dose
  Assessment of safety and tolerability of a single dose buparlisib in renal impaired subjects compared with healthy control subjects by assessing the change from baseline in ECG parameters.
Unbound plasma PK parameter AUC0-t,u | predose, 10, 30 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192, 240 hours post-dose
  Measurement of effect of renal impairment on PK of buparlisib by assessment of the PK parameters AUC0-t,u (AUC0-t,u is the area under the unbound plasma concentration-time curve from time zero to time t).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Bucharest, Romania

REFERENCES:
- See also: Results can be found for CBKM120C2113 on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14390